CLINICAL TRIAL: NCT04324866
Title: Prevalence and Incidence of COVID-19 Infection in Patients With Chronic Plaque Psoriasis on Immunosuppressant Therapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universita di Verona (Other)
Collaborators: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Paolo Gisondi, Associate Professor, Universita di Verona
Other Study IDs: Gisondi 4
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Coronavirus Infection
Keywords: psoriasis; immunosuppressant therapy; covid 19
MeSH Terms: conditions — Coronavirus Infections; Psoriasis; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nasopharyngeal swabs
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Patients with chronic plaque psoriasis on immunosuppressant therapy
  Interventions: Diagnostic Test: Nasopharyngeal swab
- Group 2: Psoriatic patients' partners
  Interventions: Diagnostic Test: Nasopharyngeal swab
- Group 3: Patients with atopic dermatitis treated with dupilumab
  Interventions: Diagnostic Test: Nasopharyngeal swab

INTERVENTIONS:
Diagnostic Test: Nasopharyngeal swab — Nasopharyngeal swab for the molecular diagnosis of COVID-19 infection

SUMMARY:
This study will assess the prevalence and incidence of COVID-19 infection in patients with chronic plaque psoriasis on immunosuppressant therapy.

DETAILED DESCRIPTION:
The ongoing COVID-19 pandemic has hit Northern Italy (including the Veneto region) particularly hard, causing several deaths and putting a huge strain on the Italian National Healthcare System. In the absence of specific treatments, preventing the infection from spreading remains the only effective measure. There is a lot of apprehension both from doctors (including dermatologists, rheumatologists and gastroenterologists) and their patients that immunosuppressive medications (biologics, methotrexate, ciclosporin and corticosteroids) might lead to an increased susceptibility to COVID-19 infection or negatively influence the course of the infection. However, there is currently a lack of scientific evidence to recommend whether immunosuppressive treatments should or should not be continued in patients who have no symptoms of COVID-19 infection. Besides, treatment discontinuation would cause flare-ups of diseases - such as plaque psoriasis, psoriatic arthritis and inflammatory bowel diseases - which are invalidating and have a relatively high prevalence in the Veneto population. In the Unit of Dermatology of the Azienda Ospedaliera Universitaria Intergrata di Verona alone, more than 2000 patients are currently being treated with immunosuppressive agents. As of now, there are no data available on the prevalence and incidence of COVID-19 infection in patients with immune-mediated diseases, nor can data from randomized clinical trials be extrapolated to the susceptibility to COVID-19 infection in patients on biologic drugs. This study aims to assess the prevalence and incidence of COVID-19 infection in patients with chronic plaque psoriasis on immunosuppressive therapy and to identify associated risk factors. Such data would prove invaluable for clinicians dealing with patients on immunosuppressive agents during the coronavirus outbreak.

ELIGIBILITY:
Group 1

Inclusion Criteria:

* Aged 18 to 75 years old
* Individuals with a clinical diagnosis of moderate-to-severe chronic plaque psoriasis confirmed by the Investigator
* Continuous immunosuppressive therapy (etanercept, adalimumab, infliximab, ustekinumab, secukinumab, ixekizumab, brodalumab, guselkumab, apremilast, methotrexate, ciclsoporin, acitretin) for the past 3 months
* Is willing and able to sign informed consent to participate

Exclusion Criteria:

* Patients unwilling to undergo noasopharyngeal swab
* Inability to give informed consent

Group 2

Inclusion Criteria:

* Aged 18 to 75 years old
* Partner of a patient with psoriasis enrolled in the study
* Is willing and able to sign informed consent to participate

Exclusion Criteria:

* Personal history of psoriasis
* Ongoing immunosuppressive therapy
* Patients unwilling to undergo noasopharyngeal swab
* Inability to give informed consent

Group 3

* Aged 18 to 75 years old
* Individuals with a clinical diagnosis of moderate-to-severe atopic dermatitis confirmed by the Investigator
* Continuous therapy with dupilumab for the past 3 months
* Is willing and able to sign informed consent to participate

Exclusion Criteria:

* Patients unwilling to undergo noasopharyngeal swab
* Inability to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll patients from the Unit of Dermatology of Azienda Ospedaliera Universitaria di Verona and their partners.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-04-01 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Point prevalence of COVID-19 infection | Baseline up to 6 months

SECONDARY OUTCOMES:
Incidence of COVID-19 infection | Baseline up to 6 months
Percentage of subjects presenting fever or respiratory symptoms | Baseline up to 6 months
Evaluate the relationship between COVID-19 infection and chronic pharmacological treatments | Baseline up to 6 months
Evaluate the relationship between COVID-19 infection and comorbid medical conditions | Baseline up to 6 months